CLINICAL TRIAL: NCT00203086
Title: A Multi-Centered, Two Arm, Open Label Extension Study (to Protocol NC-100) to Evaluate the Long-Term Safety and Efficacy of Short-Term Induction Treatment With Mitoxantrone (Novantrone®) Preceding Treatment With Glatiramer Acetate (Copaxone®) vs. Chronic Treatment With Glatiramer Acetate Alone in Relapsing Forms of Multiple Sclerosis
Brief Title: A Study to Evaluate the Long Term Safety and Effectiveness of Novantrone Therapy Followed by Copaxone Treatment for Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Siyu Liu, Vice President, North American Innovative Research & Development and Head, Teva Neuroscience
Other Study IDs: PM025
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2010-04-29 (Estimated); Status verified 2010-04

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
It is thought that treating Multiple Sclerosis with Novantrone for a short period of time prior to treatment with Copaxone may enhance the onset effect of Copaxone.

ELIGIBILITY:
Inclusion Criteria:

* Participation & completion of the NC-100 Clinical Trial.
* Able and willing to sign an Informed Consent.

Exclusion Criteria:

none

Ages: 20 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Neurology Clinics
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2005-10; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Pardo, MD, Study Director — Teva Neuroscience, Inc.